CLINICAL TRIAL: NCT02994277
Title: Pilot Study of Automatic Glycaemic Correction Systems (Closed-loop) in Patients With Type 1 Diabetes Mellitus With Continuous Subcutaneous Insulin Infusion
Brief Title: Artificial Pancreas in Latin America
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Instituto Tecnológico de Buenos Aires (Other); Universidad Nacional de La Plata (Other); Universidad Nacional de Quilmes (Unknown); University of Virginia (Other); Fundación Nuria/Cellex (Unknown)
Responsible Party: Principal Investigator, Waldo Horacio Belloso, MD, Hospital Italiano de Buenos Aires
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2680
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2017-11

CONDITIONS: Diabetes
Keywords: "Artificial Pancreas"; "control System"; "Closed loop"; diabetes; "T1DM"; "pump"; algorithm; CGM
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UVa and ITBA/UNLP algorithm arm (Experimental): To control glycaemia in T1DM patients through UVa and ITBA/UNLP algorithm
  Interventions: Device: 1° Phase: UVa algorithm 2° Phase: ITBA/UNLP algorithm

INTERVENTIONS:
Device: 1° Phase: UVa algorithm 2° Phase: ITBA/UNLP algorithm — The UVa algorithm is an already established mathematical model that can be programmed in DiAs software to manage glycaemia in T1DM through a subcutaneous insulin pump and a continous glucose monitoring. This algorthm works on a meal announcement basis and will be tested during the first phase of the trial. The ITBA/UNLP algorithm is a new development with safety mechanisms improved and without need of meal anouncement. This algorithm will be tested during the second phase of the trial.

SUMMARY:
The purpose of this study is to use closed-loop systems with the algorithms designed by the University of Virginia and by the Instituto Tecnologico de Buenos Aires (ITBA)/ Universidad Nacional de La Plata (UNLP)/ Universidad Nacional de Quilmes (UNQ) to determine the infusion of insulin in a prolonged period of time in patients with type 1 diabetes mellitus (T1DM).

DETAILED DESCRIPTION:
Aims:

1. To test University of Virginia closed-loop algorithm with meal announcement for 36 hours at our facilities.
2. To test the ability of the closed-loopInstituto Tecnologico de Buenos Aires (ITBA)/ Universidad Nacional de La Plata (UNLP)/ Universidad Nacional de Quilmes (UNQ) algorithm without meal announcement to maintain glucose control for 2 periods of 12 hours

In both cases, the adequate operation of the system will be considered verified if the system works properly at least 80% of the total connection time .

ELIGIBILITY:
Inclusion Criteria:

* Patient have been diagnosed with T1DM at least two years ago and have been using an insulin pump and a CGM for at least 6 months prior to the trial first visit.
* Patient is >18 and <65 years.
* Patient has HbA1c > 6.5 % and < 10%.
* Woman in premenopausal age agrees to use contraceptive methods.
* Woman in premenopausal age has negative B-HCG in the tests performed in the trial.
* Patient is trained in carbohydrates counting.
* Patient has signed informed consent and has the ability to understand the nature and intent of the study including the ability to comply with study procedures and is willing to keep scheduled visits.

Exclusion Criteria:

* Patient has been hospitalized for diabetic ketoacidosis in the last 12 months.
* Patient has experienced severe hypoglycemia with loss of consciousness in the last 12 months.
* Patient has a history of coronary disease or cardiac failure.
* Patient with uncontrolled arterial hypertension.
* Patient with a condition that makes the researcher believe that it might increase the chance of hypoglycemia.
* Patient has symptoms compatible with an active infectious disease.
* Patient has Cystic Fibrosis.
* Pregnant women, or women with the intention of getting pregnant; women breastfeeding.
* Patient has been hospitalized for psychiatric treatment in the last 6 months.
* Patient with a diagnosis of an adrenal disease.
* Patient has abnormal laboratory values for liver function: transaminase > 2x upper limit of normal.
* Patient has abnormal laboratory values for renal function: GFR < 60 ml/min/1.73m2
* Patient has active gastroparesis.
* Patient is under oncological treatment.
* Patient has taken acetaminophen 72 hours previous to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
System connectivity | 36 hours
  Adequate operation of the system will be considered verified if the system works properly at least 80% of the total connection time.

SECONDARY OUTCOMES:
Technical fail rate | 36 hours
Percentage of time in glycaemia between 70-180 mg/dl | 36 hours
Percentage of time in glycaemia between 181-250 mg/dl | 36 hours
Percentage of time in hypoglycaemia defined as <70 mg/dl | 36 hours
Percentage of time in hyperglycaemia defined as >180 mg/dl | 36 hours
Number of all hypoglycaemic events (syntomatic and non syntomatic) | 36 hours
Comparison of glycaemic profiles during the trial with glycaemic profiles in the days before the trial | 36 hours
Meal composition's effect in the efficacy of the system to control glycaemia | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Waldo H Belloso, MD, Study Director — Hospital Italiano de Buenos Aires

IPD SHARING:
Plan to Share IPD: No